CLINICAL TRIAL: NCT03320083
Title: Associates and Natural Course of Behavioral Insomnia of Childhood: Impact of Parent Education
Brief Title: Behavioral Insomnia of Childhood: Impact of Parent Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 09.2015.215
Record Dates: First submitted 2017-10-20; First posted 2017-10-25 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: sleep, infants, behavioural insomnia, breastfeeding
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational care derived from POSSUMS (Active Comparator): Intervention group were offered a sleep education session using behavioral change counseling communication skills, derived from the POSSUMS approach developed by Douglas P and Whittingham K. However we could not use Acceptance and Commitment Therapy (ACT), because none of the investigators had sufficient training on ACT at the time the study was conducted.
  Interventions: Behavioral: Educational care derived from POSSUMS
- Usual Care (No Intervention): General anticipatory guidance given

INTERVENTIONS:
Behavioral: Educational care derived from POSSUMS — Intervention group were offered a sleep education session on healthy practices for parent-baby sleep which included information on sleep needs, sleep hygiene, training in strategies to remove obstacles that get in the way of healthy sleep. Information were provided to guide the parent in forming an action plan based on cued care which included aligning the circadian clock with real time, removing the obstacles that get in the way of healthy sleep, physical activity, mindfulness, and relaxation techniques for mothers derived from the POSSUMS approach. However, we could not use Acceptance and Commitment Therapy, because none of the investigators had sufficient training on ACT at the time the study was conducted.
  Arms: Educational care derived from POSSUMS

SUMMARY:
Behavioral Insomnia of Childhood (BIC) is among the most prevalent problem presented to pediatricians with a reported occurrence of approximately 30% worldwide.The most widely applied treatment strategies for BIC in infants comprise behavioral procedures such as unmodified extinction; graduated extinction (ignoring the infant cries with minimal checks), or camping out. Unfortunately, breastfeeding is usually considered as an undesirable sleep association in these strategies. Moreover, less is known regarding the effects of these interventions on breastfeeding outcomes. The cued care is defined as a pattern of care characterized by sensible caregiver responsiveness, which meets the need underlying the infant's cues in a flexible manner. In this context, POSSUMS has been developed as a cued care sleep intervention, which is quite different from the conventional sleep training techniques. In the current study, investigators hypothesized that mothers receiving the cued care sleep intervention would report less sleep problems in their infants. Secondary outcomes included improvement in maternal mood and maintenance of the breastfeeding during the observation period.

DETAILED DESCRIPTION:
Behavioral Insomnia of Childhood (BIC) is among the most prevalent problem presented to pediatricians with a reported occurrence of approximately 30% worldwide.Like all the other behavioral problems, sleep problem is defined by the the parents, and influenced by parental psychopathology, parenting styles, family dynamics, culturally-based differences in values, socio-economic factors, temperament, developmental stage and medical condition of the child. Moreover, there is also data suggesting an association of depressed mood among mothers to infants with BIC. The most widely applied treatment strategies for BIC in infants comprise behavioral procedures such as unmodified extinction; graduated extinction (ignoring the infant cries with minimal checks), or camping out. The primary outcomes of these interventions include enabling infants to learn to self soothe to sleep, having less fragmented night-time sleep and longer night-time sleep periods. Unfortunately, breastfeeding is usually considered as an undesirable sleep association in these strategies. Moreover, less is known regarding the effects of these interventions on breastfeeding outcomes. Within the infant sleep research field, not breastfed but the formula fed baby is usually considered as the biological norm. However, since nursing influences both the maternal and infant sleep architecture, the outcomes of those behavioral interventions can not be accurately evaluated without considering the breastfeeding.

The cued care is defined as a pattern of care characterized by sensible caregiver responsiveness, which meets the need underlying the infant's cues in a flexible manner. In this context, POSSUMS has been developed as a cued care sleep intervention, which is quite different from the conventional sleep training techniques. This method uses the breast to make the baby go back to sleep as quickly as possible as long as the mother is happy with breastfeeding at night.

In the current study, investigators hypothesized that mothers receiving the cued care sleep intervention would report less sleep problems in their infants. Secondary outcomes included improvement in maternal mood and maintenance of the breastfeeding during the observation period.

The first part of the study was a baseline assessment of sleep problems. Software generated random number table was used to randomly allocate subjects to intervention and usual care groups. Mother-infant dyads in both groups were reassessed 3 months post intervention.

225 consecutive mother-infant dyads were assessed for eligibility at Marmara University Medical School, well- child outpatient clinic, Istanbul between 01 February 2016 and 15 April 2016. Seven did not meet the inclusion criteria, and 35 participants declined to participate. 91 were allocated to usual care, and 92 were allocated to patient education. Twenty five participants from the usual care and 1 mother infant dyad from the intervention group were lost to follow up and 157were included in the final analysis.

ELIGIBILITY:
Inclusion Criteria:

* infants' gestational age ≥37 weeks, healthy with normal birth weight (≥2.5 kg),and absence of any neonatal or postnatal medical condition

Exclusion Criteria:

* premature infants, infants with acute or chronic medical condition

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 157 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
Rates of infant sleep problems | 3 months
  Infant sleep problems reported by the mother and according to Brief Infant Sleep Questionnaire (BISQ). It is not a scale. The variables of the questionnaire included 1) nocturnal sleep duration (between the hours of 7 pm and 7 am); 2) daytime sleep duration (between the hours of 7 am and 7 pm); 3) number of night wakenings; 4) duration of wakefulness during the night hours (10 pm to 6 am); 5) nocturnal sleep-onset time (the time when the child falls asleep for the night); 6) settling time (latency to falling asleep for the night); 7) method of falling asleep; 8) location of sleep; 9) preferred body position; 10) age of child; 11) gender of child; 12) birth order; and 13) role of the responder who completed the BISQ. If the child woke up more than 3 times per night, spent more than 1 hour in wakefulness during the night, or spent less than 9 hours in sleep (day and night), then they were considered as poor sleepers

SECONDARY OUTCOMES:
Breastfeeding rates | 3 months
  Infant breastfeeding rates
Maternal depression | 3 months
  Mothers' depressive symptoms measured by Beck depression scale. The Beck depression Inventory is a 21 item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. The highest possible total score for the test is sixty three. The score between 11-16 indicates mild mood disturbance, 17-20 borderline clinical depression, 21-30 moderate depression, 31-40 severe depression, over 40 extreme depression

CONTACTS AND LOCATIONS:
Overall Officials: Perran Boran, Study Chair — Marmara University medical school